CLINICAL TRIAL: NCT04452643
Title: Prospective, Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial on the Efficacy of BACMUNE (MV130) in the Prevention of Disease Due to SARS-CoV-2 Infection in Healthcare Personnel
Brief Title: Efficacy of BACMUNE (MV130) in the Prevention of Disease Due to COVID-19 Infection in Healthcare Personnel
Acronym: Bacmune
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Not authorized by Cofepris (Mexico Competent Regulatory Authority)
Sponsor: Inmunotek S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MV130-SLG-037
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Double blind placebo control
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind placebo control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bacmune (MV130) (Active Comparator): Subject included in the active group will receive Bacmune. The dose consists on 2 spray puff every 12 hours for 45 days.
  Interventions: Biological: BACMUNE (MV130)
- Placebo (Placebo Comparator): Subject included in the placebo group will receive placebo. The dose consists on 2 spray puff every 12 hours for 45 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: BACMUNE (MV130) — BACMUNE (MV130) is a bacterial preparation that contains a mixture of Gram + and Gram - inactivated bacteria at the concentration of 300 FTU / mL (approx. 10^9 bacteria / mL)
  Arms: Bacmune (MV130)
Other: Placebo — Placebo is a solution on sodium chloride at 0.9%
  Arms: Placebo

SUMMARY:
The purpose of this trial is to assess the effect of immunotherapy with the bacterial preparation MV130 on the spread and course of SARS-CoV-2 infection in highly exposed subjets, as is the case with healthcare personnel.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, double-blind, placebo-controlled clinical trial to assess the efficacy of BACMUNE (MV130) in the prevention of disease due to SARS-VoC-2 infection in healthcare personnel

ELIGIBILITY:
Inclusion Criteria:

* Health personnel who are or have been in contact with patients with disease due to SARS-COV-2 infection within the last 14 days before randomization.
* Negative result for test against COVID-19.
* Subjects who have given informed consent.
* Men or women aged between 18 and 65 years, both included.
* Subjects who have a smartphone where they can load an APP for monitoring the symptoms.

Exclusion Criteria:

* Subjects who are participating in another clinical trial.
* Subjects who are unable to offer cooperation and/or have serious psychiatric disorders.
* Subjects who are allergic to any of the compounds included into MV130.
* Subjects who present contraindications to any of the components of BACMUNE (MV130).
* Subjects who are not able to comply with the dosage regimen.
* Subjects with immunodeficiencies.
* Subjects with malignancy involving the bone marrow or lymphoid systems.
* Pregnant or suspected pregnant women and breastfeeding women.
* Subjects in medical treatment that affects the response of the immune system. It includes corticosteroids (equal to or more than 20 mg for more than 2 weeks), immunosuppressants, biological agents (such as anti TNF-alpha monoclonal antibodies, etc.).
* Subjects with HIV.
* Subjects under treatment with metformin.
* Subjects treated with Sertraline.
* Subjects treated with statins.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of subjects with COVID-19 | 60 days
  Incidence of subjects with COVID-19, defined by the presence of:
  * Fever
  * Any of the respiratory signs and/or symptoms: cough, dyspnea, respiratory failure, runny nose/nasal obstruction.
  * Positive test for SARS-COV-2 (PCR o serology)
Severity of COVID-19 | 60 days
  Incidence of severe COVID-19, defined by CURB > 2 and/or death

SECONDARY OUTCOMES:
Seroconversion to SARS-CoV-2 | 60 days
  Rate of subjects with seroconversion to SARS-CoV-2 (negative serology at the beginning of the study and positive at the end of the study
Subjects with symptoms | 60 days
  Rate of subjects with any symptoms, whether confirmed, probable or suspected, according to the WHO definition
Hospital admission due to COVID-19 | 60 days
  The effect of the treatment on the severity of the disease will be measured based on the rate of subjects requiring hospital admission for COVID-19
Admission to an intensive care unit due to COVID-19 | 60 days
  The effect of the treatment on the severity of the disease will be measured based on the rate of subjects who require admission to an intensive care unit for COVID-19
  • Time from confirmation of SARS-CoV-2 infection to the appearance of symptoms.
Elapsed time until hospitalization | 60 days
  Elapsed time until the first symptoms of COVID-19 appears to hospitalization due to COVID-19.
Elapsed time until admission into an care unit for COVID-19 | 60 days
  Elapsed time until the first symptoms of COVID-19 appears to admission into an intensive care unit pro COVID-19.
Elapsed time until death not related to COVID-19 | 60 days
  Elapsed time until the first symptoms of COVID-19 appears to death from any cause not related to COVID-19.

CONTACTS AND LOCATIONS:
Overall Officials: Rosaura Esperanza Benitez Pérez, Principal Investigator; Felipe Monrroy López, Principal Investigator; Blanca Nohemí Zamora Mendoza, Principal Investigator
Locations (3):
- Mexico (3):
  - Instituto Nacional de Enfermedades Respiratorias (INER), Mexico City
  - Hospital General de Pachuca, Pachuca
  - Hospital de Ciudad Valles, San Luis Potosí City

IPD SHARING:
Plan to Share IPD: No